CLINICAL TRIAL: NCT04098718
Title: The Use of Benralizumab, an Interleukin-5 Receptor-α Monoclonal Antibody as Treatment of Acute Exacerbations of Airways Disease
Brief Title: Acute Exacerbations Treated With BenRAlizumab (The ABRA Study)
Acronym: ABRA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 249196; 2018-004401-79 (EudraCT Number)
Record Dates: First submitted 2019-08-09; First posted 2019-09-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2023-01

CONDITIONS: Asthma; COPD
Keywords: Exacerbations; Interleukin 5; Prednisolone; Randomised Clinical Trial
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — benralizumab; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PO open label prednisolone (in low blood eosinophils) (Other): Standard care Prednisolone 30mg given daily for 5 days to treat an exacerbation.
  Interventions: Drug: Prednisolone
- Benralizumab SC + PO placebo (Experimental): Benralizumab as a single 100mg sub cut injection and oral placebo tablet daily for 5 days
  Interventions: Drug: Benralizumab
- Benralizumab SC + PO prednisolone (Experimental): Benralizumab as a single 100mg sub cut injection and oral prednisolone 30mg daily for 5 days
  Interventions: Drug: Benralizumab; Drug: Prednisolone
- Placebo SC + PO prednisolone (Active Comparator): Placebo sub cut injection and oral prednisolone 30mg daily for 5 days.
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Benralizumab — 100mg sub cut once only
  Other Names: Fasenra
  Arms: Benralizumab SC + PO placebo; Benralizumab SC + PO prednisolone
Drug: Prednisolone — 30mg tablet daily for 5 days
  Arms: Benralizumab SC + PO prednisolone; PO open label prednisolone (in low blood eosinophils); Placebo SC + PO prednisolone

SUMMARY:
Exacerbations of asthma and COPD are an important cause of hospital admission and the main cause of annual winter bed shortages. Despite current guideline treatment with prednisolone, 40% of patients require further treatment, 15% are readmitted and, of those hospitalised, 10% die within 3 months, all by definition treatment failures. The investigators have shown that there are two dominant patterns of airway inflammation in patients presenting with an acute episode: infection associated neutrophilic airway inflammation; and non-infection related eosinophilic airway inflammation. These patterns cannot be distinguished reliably by clinical categories (i.e. asthma or COPD) or a standard clinical assessment but are identified by the peripheral blood eosinophil count. These findings raise important questions that targeted treatment based on the blood eosinophil count would result in more efficient and effective management. However, even in patients with the right pattern of airway inflammation the beneficial effects of prednisolone have to be offset against a high potential for harm, with an estimated the number needed to harm as 5 for every 10 patients treated.

Benralizumab is an interleukin-5 receptor-α monoclonal antibody, injected subcutaneously, which rapidly reduces peripheral blood eosinophils for 90 days with a satisfactory safety profile. Benralizumab treatment at stable state has been shown to increase post-bronchodilator FEV1 and reduce the rates of severe exacerbations in patients with severe eosinophilic asthma and improve lung function in patients with eosinophilic COPD. Benralizumab is an attractive candidate for the acute treatment of eosinophilic exacerbations, without the side-effects of prednisolone. The investigators propose to test the hypothesis that, for participants who have a raised eosinophil count at exacerbation, a single injection of Benralizumab alone or in combination with prednisolone will improve clinical outcomes compared to prednisolone alone. The investigators will also study the effect of prednisolone on symptoms, lung function and quality of life, in an exacerbation when the eosinophil count is not raised.

DETAILED DESCRIPTION:
Acute exacerbations of asthma and COPD are an important cause of hospital admission and the main cause of annual winter bed shortages; responsible for the majority of asthma and COPD exacerbations. Despite current guideline recommendations, treatment with oral corticosteroids (for both asthma and COPD exacerbations) and antibiotics (for COPD exacerbations) is not wholly adequate, whilst a significant number of patients suffer side effects from these medicines. Furthermore, almost 40% of patients with an exacerbation, treated in a standard way with oral prednisolone, do not respond and require further treatment or re-treatment, and depressingly following a severe COPD exacerbation, 10% die within 30 days. The risk of death in patients with asthma is especially high in those who have poorly controlled asthm5. These events are all by definition treatment failures or non-response and impact on patient outcomes. In patients with COPD the outlook is particularly bleak following a second hospital admission with a significant increase in mortality.

Inflammation in exacerbations of asthma and COPD

It is now recognised that there are two dominant patterns of airway inflammation in patients presenting with an acute wheezing illness: 1. infection associated neutrophilic airway inflammation; and 2. non-infection related eosinophilic airway inflammation; both related to asthma and COPD, with a predominance of non-infection related eosinophilic inflammation in patients with asthma. These patterns of airway inflammation are very rarely seen together and cannot be distinguished reliably by clinical categories (i.e. asthma or COPD) or a standard clinical assessment. They can however be identified by the peripheral blood eosinophil count, which is ≥2% in 90% of patients with eosinophilic airway inflammation and <2% in a similar proportion of patients with infection associated neutrophilic airway inflammation. Furthermore, these types of inflammation are consistent within patients, whether assessed when in the stable state or in the setting of an acute attack. Furthermore, patients with eosinophilic inflammation have been repeatedly shown to have more exacerbations and that incomplete suppression of eosinophilic inflammation leads to an accelerated time to next exacerbation in COPD. These findings raise important questions about our current 'one size fits all' approach to management of acute wheezing illnesses in patients with asthma and COPD and suggest that targeted treatment based on effective reduction of inflammation would result in more efficient and effective management.

Treatment of exacerbations

A key component of treatment of the acute exacerbation event in patients with asthma and COPD is systemic corticosteroids i.e. oral prednisolone often at a dose of between 30-50mg once per day for 5 to 14 days. This is especially the case in patients with eosinophilic inflammation at the onset of the exacerbation event. However, even in patients with the right pattern of airway inflammation the beneficial effects of prednisolone have to be offset against a high potential for harm. One study using systemic corticosteroids in the exacerbation setting in patients with COPD estimated the number needed to treat (NNT) to reduce 1 treatment failure episode as 10 whilst simultaneously reporting that the number needed to harm (NNH) as 5. Adverse effects include significant hyperglycaemia, leading to diabetes in approximately 8% of patients' treated; osteoporosis with recurrent prescription; and treatment induced psychosis. Moreover, in a recent retrospective analysis of hospital prescriptions for systemic corticosteroids, excluding patients with airways disease, the incidence of patients with adverse events and harm in the first 30 days of a short course prednisolone prescription was significantly high, with an incidence rate (95%CI) of sepsis of 5.3 (3.8 to 7.1); venous thromboembolism of 3.3 (2.8 to 4.0); and fracture rate of 1.9 (1.7 to 2.1). Additional difficulties with prednisolone include the short duration of action and the requirement for treatment adherence. These factors increase the chance of relapse as a result of recurrent eosinophilic airway inflammation and has been shown to be associated with an increased time to next exacerbation in a single centre study of 230 COPD patients. Alternative treatments that have a more secure, selective and prolonged beneficial effect are thus needed.

Benralizumab, an IL5 receptor alpha monoclonal antibody: benefit risk considerations and dose justification Benralizumab is a humanized afucosylated monoclonal antibody (mAb) directed towards the human interleukin-5 (IL5) alpha receptor sub-unit, found on eosinophils and basophils. Afucosylation confers enhanced antibody-dependent cellular cytotoxicity (ADCC) which results in highly efficient eosinophil depletion by apoptosis22. Single and repeated doses of benralizumab in mild to severe asthma patients' results in rapid and sustained depletion of blood eosinophils; repeat doses of benralizumab subcutaneously (SC) also markedly reduced airway mucosal/submucosal and sputum eosinophil levels. Benralizumab 30 mg SC every 8 weeks is currently approved for severe eosinophilic asthma patients age ≥ 18 whose asthma is poorly controlled by high dose ICS/LABA therapy based on 3 Phase III trials demonstrating improvements in the annual rate of asthma exacerbations, lung function, asthma symptoms, quality of life, and OCS-sparing in OCS-dependent asthma patients. More recently, the safety profile of benralizumab in severe eosinophilic asthma patients during a second year of treatment was shown to be similar to that of the first year of treatment, with no new safety concerns27.

In the only other study where single intravenous doses of benralizumab were tested vs. placebo at the time of an asthma exacerbation, the proportion of patients with at least 1 exacerbation was not different from placebo. However, benralizumab reduced asthma exacerbation rates vs. placebo by 49% (3.59 vs 1.82; P=.01) and resulting in hospitalization by 60% (1.62 vs 0.65; P=.02) and was well tolerated. This may have been influenced by i) the lack of efficacy in treating non-eosinophilic exacerbations and ii) the additional harm from prednisolone.

In a Phase 1 study in mild to moderate asthmatics with sputum eosinophilia (MI-CP166), a cohort of patients received 100 or 200 mg of benralizumab SC or placebo dosed every 4 weeks for 3 doses. In this study the incidence of all adverse events was similar between the placebo and benralizumab groups. In a Phase 2b, dose-ranging study in uncontrolled severe asthma (MI-CP220) compared the safety and efficacy of SC benralizumab at 2, 20 and 100 mg with placebo. Investigational product was dosed every 4 weeks for the first three doses and every 8 weeks for a further 4 doses. Both the benralizumab 20 mg and 100 mg treatment arms demonstrated efficacy to reduce exacerbations and improve lung function, symptoms and quality of life in patients with high blood eosinophils compared to placebo. Treatment-emergent adverse events were reported by a higher proportion of participants in the combined benralizumab groups (277 of 385, 72%) than in the placebo groups (143 of 221, 65%) and serious adverse events were reported by the same proportion of participants receiving benralizumab as for placebo at 10%.

The Phase 2a study in moderate to very severe COPD patients with sputum eosinophilia (MI-CP196) compared the safety and efficacy of benralizumab 100 mg SC to placebo dosed every 4 weeks for the first three doses and every 8 weeks for a further 5 doses. Benralizumab demonstrated numerical, albeit non-significant, improvements in acute exacerbations, lung function and quality of life in a sub-set of patients with high blood eosinophils. There was little difference between groups in the total number of treatment-emergent adverse events, the proportion of patients who reported at least one treatment-emergent adverse event, and events with an incidence of 5% or greater. A higher incidence of serious treatment-emergent adverse events were recorded in patients in the benralizumab group than in those in the placebo group (14 vs 9 patients), although none of these events were considered by the investigator to be benralizumab related.

The 100 mg SC dose of benralizumab was also extensively studied in two large Phase 3 trials32 [GALATHEA & TERRANOVA] in patients with moderate to very severe COPD. Both studies did not meet the primary endpoint of a statistically significant reduction of exacerbations. The safety and tolerability findings in the studies were consistent with those observed in previous trials with benralizumab.

Rationale for the study design

As discussed above, prednisolone is the main stay of treatment for all patients with an exacerbation of COPD. Previous work with a different IL-5 monoclonal antibody (mepolizumab) has shown efficacy in preventing COPD exacerbations in patients with a raised eosinophil count. As benralizumab is a novel agent for the treatment of COPD exacerbation, the trial will included a combination arm to assess the potential added benefit of benralizumab to prednisolone during an exacerbation of asthma and/or COPD.

Patients with asthma and/or COPD can sometimes have variable stability of their raised blood eosinophil count34. The observational arm will thus have two purposes. The first aim of the observation group will be to observe the clinical response to prednisolone when the eosinophil count in not raised and to compare this to prednisolone alone treatment when the eosinophil count is raised. It is believed and there is previous data to suggest that corticosteroids are not beneficial for patients with a low eosinophil count and may be harmful, although this remains to be the standard treatment for these patients. The second aim of the observational group will be to allow us to maintain a pool of patients who could potentially have an eosinophilic exacerbation in the future. As will be described further in this protocol, patients would be eligible to consent if they have shown a raised blood eosinophil count in the 2 years prior to consenting at Visit 1. The observational arm will capture patients who did not have a raised eosinophil count at time of their first exacerbation. They will then be allowed up to 4 non-eosinophilic exacerbations in the observational group. Patients would be unlikely to have an eosinophilic exacerbation after 4 non-eosinophilic exacerbations and therefore would not continue to be tested during further exacerbations.

Study Hypothesis

The hypothesis being tested is that for patients with an exacerbation of asthma and/or COPD, who have a raised peripheral blood eosinophil count (≥300 cells/uL), a single injection of Benralizumab alone or in combination with prednisolone, will increase the rate of recovery and reduce the rate of treatment failure, compared to prednisolone. This will also be compared this with an observational arm of prednisolone treatment (usual care) of non-eosinophilic exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give written informed consent for participation in the trial.
* Male or Female, aged ≥ 18 years or above.
* A diagnosis made in primary or secondary care, of:

  * COPD with current or historic evidence of spirometry confirming airflow obstruction (FEV1/FVC ratio <0.7) and a smoking pack year history of ≥10. Or,
  * Asthma with current or historic evidence of spirometry confirming variable airflow limitation (any one of airflow reversibility FEV1 change >200mL; and/or FEV1% change of 12%; and/or Pc20 ≤8; and/or peak flow diurnal variation; and/or variable FEV1/FVC ratio) and a smoking pack year history <10. Or;
  * COPD and asthma (as defined above)
* A history of at least 1 exacerbation requiring oral/intravenous corticosteroids in the previous 12 months.
* Prior (within 2 years) evidence of eosinophilic inflammation; including an elevated exhaled nitric oxide (FENO) ≥25ppb; and/or peripheral blood eosinophil count ≥250 cells/uL; and/or sputum eosinophils ≥3% of the total cell count.
* Female participants of child bearing potential unless surgically sterile and/or at least 2 years post-menopause must agree to use effective measures of birth control (including sexual abstinence, vasectomised sexual partner, female sterilization by tubal ligation, any effective intra-uterine device, Depo-Provera injections, oral or transdermal contraceptive) from study recruitment to 16 weeks of the last dose of IMP.
* Male participants who are sexually active with partner(s) of child-bearing potential must use an adequate method of contraception (condom) or be surgically sterile from the first dose of IMP until 16 weeks after this dose.
* In the Investigator's opinion, is able and willing to comply with all trial requirements

Exclusion Criteria:

* A known allergy to IMP (Benralizumab or prednisolone).
* Clinically important and significant pulmonary disease other than asthma or COPD (e.g. lung cancer, pulmonary fibrosis, bronchiectasis as primary respiratory problem, active pulmonary tuberculosis, cystic fibrosis, obesity hypoventilation syndrome).
* Another clinically significant pulmonary or systemic disease associated with an elevated peripheral blood eosinophil count (e.g. allergic bronchopulmonary aspergillosis, eosinophilic granulomatosis with polyangitis, hyper-eosinophilic syndrome, and helminth infection).
* Unstable ischaemic heart disease, arrhythmia, cardiomyopathy, heart failure, significant renal or hepatic impairment, uncontrolled hypertension, or ECG abnormality as defined by the investigator, which in the judgement of the investigator may put the patient at risk or negatively affect the outcome of the study.
* A confirmed (radiological) diagnosis of pneumonia 8 weeks prior to Exacerbation Visit, based on the last date of antibiotic treatment or hospitalisation date.
* An alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level that is persistently ≥1.5 times the upper limit of normal.
* Regular use of immunosuppressive medication (including but not limited to maintenance daily prednisolone (>10mg per day), hydrocortisone, azathioprine, or weekly methotrexate).
* Established use (greater than 3 months) of long-term oxygen therapy (i.e. receiving oxygen therapy for >15hours per day).
* The presence of hypercapnic ventilatory failure and/or the requirement of nocturnal non-invasive ventilation therapy.
* Scheduled elective surgery or other procedures requiring general anaesthesia during the trial.
* Participant with life expectancy of less than 6 months.
* Any other unstable significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Receipt of any licenced (e.g. omalizumab, mepolizumab or benralizumab) or other monoclonal antibody or polyclonal antibody therapy (e.g. gamma globulin) within 6 months.
* A history of known immunodeficiency disorder (including HIV-1 or HIV-2).
* Positive hepatitis B surface antigen, or positive hepatitis C virus antibody serology or a known medical history of hepatitis B or C.
* A history of drug or alcohol abuse in the previous 12 months, which in the opinion of the investigator, may compromise study data interpretation.
* A current (or within 5 years) history of solid organ or haematological malignancy.
* Female participant who is pregnant, lactating or breast-feeding.

Additional exclusion criteria on day of exacerbation (Visit 2)

* Fever recorded as >38°C measured using the tympanic temperature and/or a suspected pulmonary bacterial infection (chest radiograph demonstrating consolidation).
* Type 2 respiratory failure necessitating non-invasive or invasive ventilation
* Any clinically significant abnormal findings in physical examination, vital signs, haematology, clinical chemistry or urinalysis, which in the opinion of the investigator, may put the subject at risk because of their participation, or may influence the results of the study, or the ability to complete the duration of the study.
* An alternative cause for the increase in symptoms that are unrelated to an exacerbation such as i) suspicion or clinical evidence of pneumonia; ii) high probability and suspicion of pulmonary embolism; iii) suspicion or clinical evidence of a pneumothorax; iv) primary ischaemic event - ST or Non ST elevation myocardial infarct and left ventricular failure [i.e. not an exacerbation of asthma and/or COPD].
* Treatment with oral corticosteroids and/or hospitalisation for an exacerbation of asthma and/or COPD in the previous 4 weeks prior to randomisation.
* More than 12 hours of oral corticosteroid treatment for a current exacerbation
* Pregnancy or a positive urinary βHCG
* Donation of blood, plasma or platelets within 90 days prior to Visit 2.
* Receipt of blood products within 30 days prior to Visit 2.
* Participants who have participated in another research trial involving an investigational product in the past 4 weeks or 5 half-lives prior to visit 2
* Treatment with allergy immunotherapy, actively or within 90 days prior to Visit 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2021-03-29 (Actual); Primary Completion 2024-02-19 (Estimated); Study Completion 2024-11-19 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in respiratory visual analogue scale symptom scores with Benralizumab treatment with and without prednisolone | Day 0 to 28
  Visual analogue scale (VAS) symptom score. 0-100 mm. Patient marks how well they feel. Result reported in millimetres. A higher score reflects worse symptoms. 5 subscales of 0-100mm will be used. The 5 subscales will assess breathlessness, cough, wheeze, sputum volume and sputum production. Subscales will be summed and total score for each day will be analysed.
Rate of treatment non response with Benralizumab treatment with and without prednisolone | Day 7
  Rate of treatment non response will be defined as as a composite end-point of i) worsening of symptoms which require further treatment or hospitalisation requiring the need of systemic corticosteroids and ii) death from any cause within 90 days of randomisation.
Rate of treatment non response with Benralizumab treatment with and without prednisolone | Day 28
  Rate of treatment non response will be defined as as a composite end-point of i) worsening of symptoms which require further treatment or hospitalisation requiring the need of systemic corticosteroids and ii) death from any cause within 90 days of randomisation.
Rate of treatment non response with Benralizumab treatment with and without prednisolone | Day 90
  Rate of treatment non response will be defined as as a composite end-point of i) worsening of symptoms which require further treatment or hospitalisation requiring the need of systemic corticosteroids and ii) death from any cause within 90 days of randomisation.

SECONDARY OUTCOMES:
Evaluate the effect of Benralizumab on time to next exacerbation | Day 28, 90 and 360
  Time to next exacerbation
Evaluate the effect of Benralizumab on quality of life questionnaire | Day 0, 7, 14, 28 and 90
  European Quality of Life-5 dimension-3 level (EQ 5D 3L) questionnaire. A higher number on each of the 5 dimension reflects worse quality of life
Evaluate the effect of Benralizumab on breathlessness | Day 0, 7, 14, 28 and 90
  Medical Research Council (MRC) breathlessness score. A higher score reflects worse breathlessness
Evaluate the effect of Benralizumab on COPD Assessment Test (CAT) | Day 0, 7, 14, 28 and 90
  CAT questionnaire. A higher score (max score of 40) reflects worse COPD symptoms
Evaluate the effect of Benralizumab on asthma control questionnaire (ACQ-6) | Day 0, 7, 14, 28 and 90
  ACQ-6. Result reported as average of 6 questions. Result range 0-6. Higher result reflects worse asthma control
Evaluate the effect of Benralizumab on asthma quality of life questionnaire (AQLQ) | Day 0, 7, 14, 28 and 90
  AQLQ. 32 item questionnaire with each item rated 0 to 7 on a Likert Scale. A higher score reflects better asthma related quality of life.
Evaluate the effect of Benralizumab on asthma control test (ACT) questionnaire | Day 0, 7, 14, 28 and 90
  ACT questionnaire. 5 point questionnaire. Likert scale of 1-5 for each item. Score range 5-25. Higher score reflects better asthma control
Evaluate the effect of Benralizumab on spirometry | Day 0, 7, 14, 28 and 90
  Forced expiratory volume in 1 second (in litres). Greater volume reflects better lung function.
Evaluate the effect of prednisolone on respiratory symptoms | Day 0 and 28
  Visual analogue scale (VAS) symptom score. 0-100 mm. Patient marks how well they feel. Result reported in millimetres. A higher score reports fewer symptoms.
Evaluate the effect of prednisolone on rates of treatment non response | Day 7 and 28
  Rates of treatment non response
Evaluate the effect of prednisolone on time to next exacerbation | Day 28 and 90
  Time to next exacerbation
Evaluate the effect of prednisolone on on quality of life questionnaire | Day 0, 7, 14 and 28
  European Quality of Life-5 dimension-3 level (EQ 5D 3L) questionnaire. A higher number on each of the 5 dimension reflects worse quality of life
Evaluate the effect of prednisolone on breathlessness | Day 0, 7, 14 and 28
  Medical Research Council (MRC) breathlessness score. A higher score reflects worse breathlessness
Evaluate the effect of prednisolone on COPD Assessment Test | Day 0, 7, 14 and 28
  CAT questionnaire. A higher score (max score of 40) reflects worse COPD symptoms
Evaluate the effect of prednisolone on asthma control questionnaire (ACQ-6) | Day 0, 7, 14 and 28
  ACQ-6. Result reported as average of 6 questions. Result range 0-6. Higher result reflects worse asthma control
Evaluate the effect of prednisolone on asthma quality of life questionnaire (AQLQ) | Day 0, 7, 14 and 28
  AQLQ. 32 item questionnaire with each item rated 0 to 7 on a Likert Scale. A higher score reflects better asthma related quality of life.
Evaluate the effect of prednisolone on Asthma control test (ACT) questionnaire | Day 0, 7, 14 and 28
  ACT questionnaire. 5 point questionnaire. Likert scale of 1-5 for each item. Score range 5-25. Higher score reflects better asthma control
Evaluate the effect of prednisolone on spirometry | Day 0, 7, 14 and 28
  Forced expiratory volume in 1 second (in litres). Greater volume reflects better lung function

OTHER OUTCOMES:
Sputum eosinophil count | Day 0, 7, 14, 28 and 90.
  Sputum eosinophil count (data reported as number of eosinophils and proportion of eosinophils as a proportion of 400 non squamous cells seen on microscopy
Sputum neutrophil count | Day 0, 7, 14, 28 and 90.
  Sputum neutrophil count (data reported as number of neutrophils and proportion of neutrophils as a proportion of 400 non squamous cells seen on microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Mona Bafadhel, PhD, MBChB, Principal Investigator — Nuffield Department of Medicine, University of Oxford, UK
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramakrishnan S, Russell REK, Mahmood HR, Krassowska K, Melhorn J, Mwasuku C, Pavord ID, Bermejo-Sanchez L, Howell I, Mahdi M, Peterson S, Bengtsson T, Bafadhel M. Treating eosinophilic exacerbations of asthma and COPD with benralizumab (ABRA): a double-blind, double-dummy, active placebo-controlled randomised trial. Lancet Respir Med. 2025 Jan;13(1):59-68. doi: 10.1016/S2213-2600(24)00299-6. Epub 2024 Nov 29. PMID 39615502